CLINICAL TRIAL: NCT06567015
Title: Phase I/II First-In-Human Open-label Trial to Assess Safety and Efficacy of STX-241 in Participants With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) Resistant to EGFR Tyrosine Kinase Inhibitors (TKIs).
Brief Title: Study of FIH of STX-241 in Locally Advanced or Metastatic NSCLC Resistant to EGFR TKIs
Acronym: STX-241 FIH
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: F60087CI101; 2023-510203-21-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-03; First posted 2024-08-22 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- STX-241/PFL-241 (Experimental): Part 1: Dose Escalation and Backfilling components (Phase Ia) Participants will receive oral (PO) STX-241/PFL-241 twice daily (BID) at fixed doses: 10 mg, 20 mg, 40 mg, 80 mg, 120 mg, 180 mg on a continuous dosing schedule
  Part 2: Dose Range Optimization (Phase Ib). Participants will receive oral (PO) STX-241/PFL-241 twice daily (BID) at fixed doses selected from Part 1 within the OBD-MTD range for Part 2 on a continuous dosing schedule.
  Interventions: Drug: STX-241

INTERVENTIONS:
Drug: STX-241 — Film-coated tablet
  Route of administration: Oral
  Other Names: PFL-241

SUMMARY:
The goal of this First-In-Human (FIH) Phase I/II trial is to establish the safety profile, determine the Recommended Phase II Dose (RP2D), explore the pharmacokinetic (PK) exposure and pharmacodynamic (PD) properties as well as assess the efficacy of STX-241/PFL-241, a mutant selective Central Nervous System (CNS)-penetrant fourth generation EGFR TKI, in participants with locally advanced or metastatic NSCLC that progressed during or following third generation EGFR TKI such as osimertinib due to C797X double acquired (secondary) mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent for participation in the trial obtained according to International Council for Harmonisation of Technical Requirements of Pharmaceuticals for Human Use (ICH) Good Clinical Practice (GCP), and national/local regulations.
2. Male or female ≥ 18 years of age at the time of signing informed consent.
3. Histological confirmation of locally advanced or metastatic, EGFR-mutant (ex19del or L858R mutations) non-small cell lung cancer (NSCLC) Stage IIIB/C or IV (AJCC 8th edition) not eligible for curative intent surgery or chemoradiation.
4. Part 1&2 Disease progression on a 3rd generation EGFR TKI-based therapy (monotherapy or in combination) received at any prior line of treatment.
5. Tumor mutation profile:

   • Part 1 (backfilling component) and Part 2: Presence of C797X and absence of T790M mutations documented locally (as part of clinical practice) on a sample (blood or tissue) collected after progression on treatment with 3rd generation EGFR TKI.
6. Part 1 (Backfilling component), Part 2: At least one measurable target lesion according to RECIST v1.1.
7. Eastern cooperative oncology group (ECOG) performance status 0-1.
8. Adequate organ function as defined below:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
   * Platelets ≥ 75 x 10^9/L
   * Hemoglobin ≥ 90 g/L.
   * Serum total bilirubin ≤ 1.5 x ULN or ≤ 3.0 × ULN for participants with documented Gilbert's syndrome.
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 x ULN. If the participant has liver metastases, AST and ALT ≤5 × ULN.
   * Estimated glomerular filtration rate (GFR) ≥ 50 mL/min by CKD-EPI equation
9. Adequate cardiac function as defined below:

   * Mean QT interval corrected for heart rate according to Fridericia's formula (QTcF) value ≤ 470 msec for women and ≤ 450 msec for men and no history of long QT syndrome or risk factors for torsade de pointe.
   * Left ventricular ejection fraction (LVEF) ≥ 50% .
   * Systolic blood pressure < 150 mmHg and diastolic blood pressure < 100 mmHg
10. Female participants of childbearing potential:

    * Negative highly sensitive serum β-HCG test performed within 7 days prior to first dose of STX-241 (C1D1) and a negative urine pregnancy test performed prior to C1D1.
    * Agreement to use one highly effective contraceptive method (as defined in protocol and according to local regulations), starting at screening period, throughout the trial and until at least 182 days (i.e. more than 5 estimated STX- 241 half-lives (2 days) plus 6 months (180 days)) after the last dose of STX-241. If the highly effective method of contraception is a hormonal contraceptive method, it must be supplemented by one additional effective (barrier) method of contraception.
    * Agreement to not donate eggs (ova, oocytes) for the purpose of assisted reproduction during the trial and for a period of 182 days after the last dose of STX-241.

    Note: a female participant of childbearing potential is a woman who is not permanently sterilized or not postmenopausal (postmenopausal is defined as 12 months with no menses without an alternative medical cause).
11. Male participants/partners with female spouse/partners of childbearing potential must agree to take appropriate precautions to avoid fathering a child, i.e.:

    * Consistently use a barrier method [e.g., condom with spermicidal foam / gel / film /cream/suppository], and his female partner use a highly effective method of contraception as defined in protocol and according to local regulations), starting at screening and continuing throughout the trial period and for 92 days (ie. more than 5 estimated STX-241 half-lives (2 days) plus 3 months (90 days)) after the last dose of STX-241.
    * Not donate sperm from Day 1 (first administration of STX-241) until at least 92 days after the last dose of STX-241.

NOTE: Other protocol defined inclusion criteria may apply.

Exclusion Criteria:

1. Participant candidate for targeted therapies available to them (such as but not limited to therapies targeting ALK, BRAF, MET, NTRK, ROS1) as identified by local testing performed after progression to the last line of systemic therapy.
2. Participant with rapid progressive disease eligible to receive a platinum-based chemotherapy.
3. Participant unable ingest or digest tablets. This can be caused by any impaired gastrointestinal function or disease, such as for example: ulcerative diseases, malabsorption syndrome, small bowel resection, ileus, etc. or any condition causing uncontrolled nausea, vomiting or diarrhea.
4. History of a primary malignancy other than NSCLC with the exception of:

   * Participants with a previous malignancy that completed all anticancer treatment at least 2 years before signing informed consent and with no evidence of residual disease from the prior malignancy at screening.
   * Malignancies with a negligible risk of metastasis or death (i.e. 5-year overall survival rate > 90%) that are adequately treated - Examples include, but are not limited to, completely resected basal cell carcinoma and squamous cell carcinoma of skin, melanoma in situ, curatively treated prostate cancer, breast cancer and early gastric cancer cured by endoscopic mucosal resection or endoscopic submucosal dissection.
5. Spinal cord compression or CNS metastases that are associated with progressive neurological symptoms or require increasing doses of corticosteroids to control the CNS disease. If a participant requires corticosteroids for management of CNS disease, the dose must have been stable for 2 weeks prior to enrollment in the trial.
6. History of hypersensitivity to active or inactive ingredients of STX-241, or drugs with a similar chemical structure or from the same class.
7. Active, bacterial, fungal, or viral infection, including, but not limited to: Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), and known Human Immunodeficiency Virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS)-related illness, tuberculosis or an infection requiring systemic therapeutic treatment within 2 weeks prior to Day 1 (first administration of STX-241).

   Note: Participants with known HIV infection are permitted if they have controlled infection (undetectable viral load [HIV ribonucleic acid polymerase chain reaction (PCR)] and CD4 count >350 either spontaneously or on a stable antiviral regimen). For participants with controlled HIV infection, monitoring will be performed per local standards.
8. Positive SARs-CoV-2 or variants of SARs-CoV2 RT-PCR test or suspected to be infected with SARs-CoV2 or variants of SARsCoV2 with confirmation pending within 2 weeks of first dose of STX-241.
9. Impaired cardiovascular function or clinically significant cardiovascular disease (either active or within 6 months prior to signing informed consent), including any of the following:

   * Myocardial infarction, acute coronary syndromes including unstable angina, coronary/peripheral artery bypass graft, coronary angioplasty or stenting.
   * Symptomatic congestive heart failure (New York Heart Association Classification Class ≥ II).
   * Cerebrovascular accident or transient ischemic attack.
   * Symptomatic bradycardia, requirement for anti-arrhythmic medication.
   * Ongoing cardiac dysrhythmias of NCI-CTCAE Grade ≥2.
10. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection or psychiatric illness/social situation that would limit compliance with trial requirements.
11. Past medical history of Interstitial Lung Disease (ILD), drug-induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD.
12. Past medical history of Stevens-Jonhson Syndrome (SJS) or Toxic epidermal necrolysis (TEN) or any evidence of clinically active SJS/TEN.
13. Women who are breast feeding.
14. Prior anticancer therapy:

    * EGFR-targeted TKI within 7 days prior to the first dose of STX-241.
    * Any other systemic anticancer therapy within 28 days or 5 half-lives prior to the first dose of STX-241, whichever is the shortest, but with a minimum of 14 days in all circumstances.
    * Radiotherapy to a large field or including a vital organ (including whole brain radiotherapy or stereotactic radiosurgery to brain) within 14 days before the first dose of STX-241.
15. Live attenuated vaccine received within 30 days prior to the first dose of STX-241.
16. Any toxicities from prior therapy with a NCI-CTCAE Grade ≥1 at the time of the first dose of STX-241 (C1D1). Exceptions include alopecia (any grade), fatigue with a Grade ≤2, and peripheral neuropathy with a Grade ≤2.
17. Major surgical procedure within 14 days of the first dose of STX-241 (procedures such as central venous catheter placement, tumor needle biopsy, and feeding tube placement are not considered major surgical procedures). Sequelae of surgical procedures must have resolved, including adequate wound healing, prior to the first dose of STX-241.
18. Treatment with a prohibited medication or herbal remedy known to be strong CYP1A2 or CYP3A4 inducers, strong CYP1A2 or CYP3A4 inhibitors, sensitive CYP1A2, CYP2B6 and CYP3A4 substrates, sensitive MATE1 and OATP1B1 substrates and proton pump inhibitors (PPI) and H2 antagonists unless discontinued prior to the first administration of STX-241 within the following timeframe:

    * At least 5 half-lives plus 14 days for strong CYP inducers.
    * At least 5 half-lives for CYP inhibitors, CYP/transporter substrates, proton pump inhibitor (PPI) and H2 antagonists.
19. Participation in a clinical trial with administration of an investigational drug within 5 half-lives plus 14 days of the investigational drug, before the first dose of STX-241.
20. Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e. g, could compromise the participant's well-being) or would prevent, limit, or confound the protocol-specified assessments.
21. Employee or family member of the investigator or site staff.

NOTE: Other protocol defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2027-11-20 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Safety: Part 1 and Part 2: Safety: Incidence and severity of treatment emergent adverse events (TEAEs)/serious adverse events (SAEs), according to NCI-CTCAE v5.0 criteria. | Screening to Safety Follow-up (30 days post last dose)
Part 1 and Part 2: Tolerability: Incidence of TEAEs/SAEs leading to STX-241 dose reductions, interruptions or discontinuations. | Screening to Safety Follow-up (30 days post last dose)
Part 1: Maximum Tolerated Dose (MTD): Incidence of Dose-Limiting Toxicities (DLTs) | From first STX-241 intake until 28 days post first dose (28 days post first dose)
Part 1: Optimal Biologically Active Dose (OBD) | From the first STX-241 intake up to 24 months
Part 2: Recommended Phase II Dose (RP2D) of STX-241 | From the first STX-241 intake up to 24 months
Part 2: cORR (Confirmed Overall Response Rate) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 per investigator. | Up to 24 months

SECONDARY OUTCOMES:
All Parts: PK exposure parameter: Maximum Plasma Concentration (Cmax) | Part 1 and Part 2: C1 Day 1, Day 2, Day 15; C2 Day 1; C3 Day 1; - each cycle is 28 days
All Parts: PK exposure parameter: Time To Maximum Plasma Concentration (Tmax) | Part 1 and Part 2: C1 Day 1, Day 2, Day 15; C2 Day 1; C3 Day 1; - each cycle is 28 days
All Parts: PK exposure parameter: Area Under The Plasma Concentration-Time Curve From Time Zero To Dosing Interval (AUC0-tau) | Part 1 and Part 2: C1 Day 1, Day 2, Day 15; C2 Day 1; C3 Day 1; - each cycle is 28 days
All Parts: PK exposure parameter: Area Under The Plasma Concentration-Time Curve From Time Zero To Time With Last Measurable Concentration (AUC0-t) | Part 1 and Part 2: C1 Day 1, Day 2, Day 15; C2 Day 1; C3 Day 1; - each cycle is 28 days
All Parts: PK exposure parameter: Area Under The Plasma Concentration-Time Curve From Time Zero To Infinity (AUC0-∞) | Part 1 and Part 2: C1 Day 1, Day 2, Day 15; C2 Day 1; C3 Day 1; - each cycle is 28 days
All Parts: PK exposure parameter: Terminal Elimination Half-Life (t½) | Part 1 and Part 2: C1 Day 1, Day 2, Day 15; C2 Day 1; C3 Day 1; - each cycle is 28 days
All Parts: PK exposure parameter: Apparent Terminal Elimination Rate Constant (λz) | Part 1 and Part 2: C1 Day 1, Day 2, Day 15; C2 Day 1; C3 Day 1; - each cycle is 28 days
All Parts: PK exposure parameter: Apparent Clearance (CL/F) | Part 1 and Part 2: C1 Day 1, Day 2, Day 15; C2 Day 1; C3 Day 1; - each cycle is 28 days
All Parts: PK exposure parameter: Apparent Volume Of Distribution (Vz/F) | Part 1 and Part 2: C1 Day 1, Day 2, Day 15; C2 Day 1; C3 Day 1; - each cycle is 28 days
All Parts: PK exposure parameter: Peak Plasma Concentration (Cmax) | Part 1 and Part 2: C1 Day 1, Day 2, Day 15; C2 Day 1; C3 Day 1; - each cycle is 28 days
All Parts: PK exposure parameter: Area Under The Plasma Concentration versus Time Curve (AUC) | Part 1 and Part 2: C1 Day 1, Day 2, Day 15; C2 Day 1; C3 Day 1; - each cycle is 28 days
All Parts: PK exposure parameter: Trough Plasma Concentration (Ctrough) | Part 1 and Part 2: C1 Day 1, Day 2, Day 15; C2 Day 1; C3 Day 1; - each cycle is 28 days
Part 1: cORR by Investigator Review (IR) in accordance to RECIST version 1.1. | Up to 24 months
All parts: DCR (Disease Control Rate) by IR in accordance to RECIST version 1.1. | Up to 24 months
All parts: TTR (Time To Response) by IR in accordance to (RECIST version 1.1. | Up to 24 months
All parts: DOR (Duration of Response) by IR in accordance to RECIST version 1.1. | Up to 24 months
Part 2: PFS (Progression-Free Survival) ( by IR in accordance to RECIST version 1.1. | Up to 24 months
Part 2: Overall Survival | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (16):
- United States (2):
  - Sarah Cannon Research Institute (SCRI) (The SCRI Oncology Research Consortium), Nashville, Tennessee
  - Oncology Consultants (OC) - Texas Medical Center - Cancer Center, Houston, Texas
- China (2):
  - Shanghai East Hospital, Tongji University, Shanghai
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
- France (5):
  - Centre Léon Bérard, Lyon
  - CHU Hôpital de la Timone, Marseille
  - Institut de Cancérologie de l'Ouest (ICO) - René Gauducheau, Saint-Herblain
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Universitätsklinikum Carl Gustav Carus Dresden, Dresden, Germany
- Netherlands Cancer Institute, Amsterdam, Netherlands
- Spain (3):
  - Vall d'Hebron Institut d'Oncologia, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Centro Integral Oncológico Clara Campal (CIOCC), Madrid
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pierre Fabre is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies as defined in our commitments. These requests are reviewed and approved by an independent review panel on the basis of scientific ground. All data provided if any is anonymized to respect the privacy of trial participants in line with applicable laws and regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: This trial data availability is according to the criteria and process described in our website
URL: https://clinicaltrials.pierre-fabre.com/en/our-commitments

REFERENCES:
- See also: For eligible studies, qualified researchers may request access to individual patient level clinical data. See Pierre Fabre's commitment to transparency of clinical study information Pillar 5. — https://clinicaltrials.pierre-fabre.com/en/our-commitments